CLINICAL TRIAL: NCT05271552
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Efficacy And Safety Study of PRN Dosing of BXCL501 Over A 12 Week Period In Subjects With Agitation Associated With Dementia
Brief Title: Dexmedetomidine in the Treatment of Agitation Associated With Dementia (TRANQUILITY II)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioXcel Therapeutics Inc (Industry)
Collaborators: Cognitive Research Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BXCL501-303
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Results first posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Agitation; Dementia
MeSH Terms: conditions — Psychomotor Agitation; Dementia | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double-Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1- 40 Micrograms (Experimental): Sublingual film containing 40 Micrograms Dexmedetomidine
  Interventions: Drug: BXCL501
- Cohort 2- 60 Micrograms (Experimental): Sublingual film containing 60 Micrograms Dexmedetomidine
  Interventions: Drug: BXCL501
- Placebo (Placebo Comparator): Sublingual Placebo film
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: BXCL501 — Sublingual Film
  Other Names: Dexmedetomidine
  Arms: Cohort 1- 40 Micrograms; Cohort 2- 60 Micrograms
Drug: Matching Placebo — Sublingual Placebo Film
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
A study to determine the safety and efficacy of BXCL501 dosing for episodes of agitation associated with dementia when they occur (given as needed [PRN]), for a maximum of 28 doses within a 12-week treatment period.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled, parallel group, 3-arm study assessing efficacy, safety, and tolerability of two doses of BXCL501 in male and female subjects (65 years and older) with acute psychomotor agitation. Subjects will be dosed PRN with a maximum of 28 doses over a 12-week period. Once a subject has received 28 doses of BXCL501, they will continue to be followed for the remainder of the 12-week study period.

Approximately 150 subjects will participate in this study. Subjects will receive a single film consisting of BXCL501 40 µg dose or BXCL501 60 µg dose or placebo in a 1:1:1 randomization scheme. Subjects must reside in a care facility where all study-related procedures and study drug dosing will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects must have a diagnosis of probable AD based on NIA-AA criteria (2018)
2. Episodes of psychomotor agitation (e.g., kick, bite, flailing)
3. Subjects exhibit behaviors that are congruent with the International Psychogeriatric Association criterion for agitation representing a change from the subject's usual behavior
4. A score of 15 to 23 on the Mini-Mental State Exam (MMSE)
5. Subjects who read, understand, and provide written informed consent, or who have a LAR to provide consent on their behalf
6. Subjects who are deemed to be medically appropriate for study participation by the principal investigator
7. Participants who agree to use a medically acceptable and effective birth control method

Exclusion Criteria:

1. Subjects with dementia or other memory impairment not due to probable AD.
2. Clinical diagnosis of probable AD should not be applied when there is evidence of a cerebrovascular incident temporally related to the worsening of cognitive function.
3. Subjects with agitation caused by acute intoxication.
4. Subjects with significant risk of suicide or homicide per the investigator's assessment.
5. Subjects who are medically unstable or in recovery. Note: Subjects with a remote (>5 years) history of stroke may be included, regardless of size/location.
6. History of clinically significant syncope or syncopal attacks, orthostatic hypotension within the past 2 years, current evidence of hypovolemia, orthostatic hypotension, bradycardia.
7. Subjects who had a total score of >13 (ie, high fall risk) on the John Hopkins Fall Risk Assessment Tool.
8. Subjects with laboratory or ECG abnormalities.
9. Subjects who have received an investigational drug within 30 days prior to Screening.
10. Subjects who are currently suffering from substance abuse. Patients with a potential cause for delirium (relatively recent onset agitation and dementia)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 151 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Risinger, MD, Study Chair — BioXcel Therapeutics
Locations (11):
- United States (11):
  - BioXcel Clinical Research Site, Phoenix, Arizona
  - BioXcel Clinical Research Site, Long Beach, California
  - BioXcel Clinical Research Site, Daytona Beach, Florida
  - BioXcel Clinical Research Site, Lady Lake, Florida
  - BioXcel Clinical Research Site, Maitland, Florida
  - BioXcel Clinical Research Site, Miami Lakes, Florida
  - BioXcel Clinical Research Site, North Miami, Florida
  - BioXcel Clinical Research Site, Marrero, Louisiana
  - BioXcel Clinical Research Site, Springfield, Massachusetts
  - BioXcel Clinical Research Site, Berlin, New Jersey
  - BioXcel Clinical Research Site, Toms River, New Jersey

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in United States from 18 April 2022 to 21 April 2023.
Period: Overall Study
Arm/Group | Cohort 1- 40 Micrograms | Cohort 2- 60 Micrograms | Placebo
Started | 48 | 50 | 53
Completed | 38 | 29 | 32
Not Completed | 10 | 21 | 21
Not completed — Adverse Event | 4 | 6 | 3
Not completed — Death | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 5 | 4
Not completed — Withdrawal by Subject | 0 | 4 | 7
Not completed — Other medical reason. | 1 | 2 | 0
Not completed — Other | 3 | 3 | 6

BASELINE CHARACTERISTICS:
Population: The Safety Population includes all subjects who received the study treatment. Two subjects randomized to Placebo voluntarily withdrew before dosed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1- 40 Micrograms | Cohort 2- 60 Micrograms | Placebo | Total
Number analyzed (Participants) | 48 | 50 | 51 | 149
Age, Continuous [Mean (Standard Deviation); unit: Years] | 79.4 (6.44) | 79.5 (8.14) | 80.0 (7.48) | 79.6 (7.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 30 | 33 | 90
  Male | 21 | 20 | 18 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 22 | 19 | 59
  Not Hispanic or Latino | 30 | 28 | 32 | 90
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 13 | 5 | 11 | 29
  White | 35 | 43 | 39 | 117
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2
Baseline Positive and Negative Syndrome Scale - Excited Component (PEC) [Mean (Standard Deviation); unit: units on a scale] — The scale is 5 - 35, with the higher number presenting the worse outcome. Each of the sub scales is on the scale of 1 - 7 and the sub scales are summed to obtain PEC. The sub scales are the following items from PANSS: hostility, uncooperativeness, tension, poor impulse control, and excitement.
  units on a scale | 17.3 (2.18) | 18.0 (2.26) | 17.5 (2.62) | 17.6 (2.36)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Positive and Negative Syndrome Scale- Excited Component (PEC) Total Score for the First Episode of Agitation
Description: The Positive and Negative Syndrome Scale - Excited Component (PEC) comprises 5 items associated with agitation: poor impulse control, tension, hostility, uncooperativeness, and excitement; each scored 1 (minimum) to 7 (maximum). The PEC, the sum of these 5 subscales, thus ranges from 5 (absence of agitation) to 35 (extremely severe)
Time Frame: 120 minutes
Population: Full analysis set included all subjects who took any study medication and who had both baseline and at least one efficacy assessment after dosing.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cohort 1- 40 Micrograms | Cohort 2- 60 Micrograms | Placebo
Number analyzed (Participants) | 48 | 50 | 51
score on a scale | -5.7 (0.6) | -7.5 (0.6) | -5.4 (0.6)

2. Secondary Outcome: Absolute Change From Baseline in Positive and Negative Syndrome Scale- Excited for the First Episode of Agitation
Description: as for outcome 1
Time Frame: 30 minutes
Population: Full Analysis Set (FAS) included all subjects who took any study medication and who had both baseline and at least one efficacy assessment after dosing.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cohort 1- 40 Micrograms | Cohort 2- 60 Micrograms | Placebo
Number analyzed (Participants) | 48 | 50 | 51
score on a scale | -2.5 (0.5) | -3.6 (0.5) | -3.4 (0.5)

3. Secondary Outcome: Absolute Change From Baseline in Positive and Negative Syndrome Scale- Excited for the First Episode of Agitation
Description: as for outcome 1
Time Frame: 60 minutes
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cohort 1- 40 Micrograms | Cohort 2- 60 Micrograms | Placebo
Number analyzed (Participants) | 48 | 50 | 51
score on a scale | -4.2 (0.6) | -6.2 (0.6) | -4.2 (0.6)

4. Secondary Outcome: Absolute Change From Baseline in Positive and Negative Syndrome Scale- Excited for All Episodes of Agitation
Description: as for outcome 1
Time Frame: 120 minutes
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Cohort 1- 40 Micrograms | Cohort 2- 60 Micrograms | Placebo
Number analyzed (Participants) | 48 | 50 | 51
score on a scale | -5.8 (0.5) | -7.4 (0.5) | -5.2 (0.5)

ADVERSE EVENTS:
Time Frame: 24 hours after dose administration (treatment emergent adverse events)
Description: The AEs are summarized as treatment emergent adverse events which started within 24 hours after any dose. Subjects are counted once at the highest severity at each organ class and preferred term. The terms were coded using MedDRA, Version 25.0.
Arm/Group | Cohort 1- 40 Micrograms | Cohort 2- 60 Micrograms | Placebo
All-Cause Mortality (participants affected / at risk) | 1/48 | 1/50 | 1/51
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/50 | 0/51
Other Adverse Events (participants affected / at risk) | 6/48 | 16/50 | 2/51
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1- 40 Micrograms (N=48) | Cohort 2- 60 Micrograms (N=50) | Placebo (N=51)
Somnolence (Nervous system disorders) | 2 | 3 | 0
Hypotension (Vascular disorders) | 0 | 3 | 0
Orthostatic Hypotension (Vascular disorders) | 2 | 2 | 0
Bradycardia (Cardiac disorders) | 1 | 2 | 0
Lethargy (Nervous system disorders) | 1 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fracture treatment (Surgical and medical procedures) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
"Principal Investigator and Institution may not use it for any publication, presentation, disclosure, or commercial purposes (i.e., furtherance of the interest of any profit-making enterprise). Methods, assessments or procedures used in the collection of the Data, as well as the Study Drug name, Sponsor name and protocol title, are considered confidential and may not be disclosed for scientific, educational or other purposes as specified in paragraph 6."

DOCUMENTS (2):
  • Study Protocol (2022-11-18): https://cdn.clinicaltrials.gov/large-docs/52/NCT05271552/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-17): https://cdn.clinicaltrials.gov/large-docs/52/NCT05271552/SAP_001.pdf